CLINICAL TRIAL: NCT02837107
Title: Study of Supplement's Antioxidant Properties That Contains Natural Extracts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Elizabeth Fragopoulou, Assistant Professor of Biological Chemistry, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HAROKOPIO UNIVERSITY
Record Dates: First submitted 2016-05-23; First posted 2016-07-19 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Supplement (Active Comparator): The supplement (Mind Master) were custom prepared and donated by LR Healthy and Beauty Systems LTD. The supplement contained per 80ml, aloe barbadensis miller gel (USA/Mexico 36%), grape juice, Polygonum cuspidatum extract (that contain 10% resveratrol), green tea extract, 1.1 mg vitamin B1 (100% RDA), 2.5 µg vitamin B12 (100% RDA), 12 mg vitamin E (α - ΤΕ) (100% RDA), coenzyme Q10, 200 µg folic acid (100% RDA), ascorbic acid, 27.5 µg selenium (100% RDA), 4.2 mg iron (100% RDA).
  Interventions: Dietary Supplement: Mind Master
- Placebo (Placebo Comparator): A look-alike placebo were prepared and donated by LR Healthy and Beauty Systems LTD. The placebo contained Aloe barbadensis Miller Gel (USA/Mexico 3.6%), ascorbic acid, and some excipients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mind Master — 80ml Mind Master / day for 8 weeks
  Other Names: Mind Master LR Health & Beauty Systems
  Arms: Supplement
Dietary Supplement: Placebo — 80ml a look-alike Placebo / day for 8 weeks
  Arms: Placebo

SUMMARY:
While it is well accepted that a low level of RONS production is necessary to maintain physiological function, too much formation of RONS are believed to participate in biomolecules damage. Damage of lipids, proteins and DNA/RNA, to cellular and tissue level, as a consequence of oxidative stress has been linked to a number of serious diseases, including cancer, cardiovascular diseases (CVDs) such as hypertension and atherosclerosis, neurodegenerative diseases such as Parkinson's disease and Alzheimer's dementias, diabetes and the process of aging.

The dietary intake of antioxidants is thought to play a major role in oxidative stress network. Many epidemiologic studies have reported an inverse association between vegetable and fruit consumption with reduced risk of chronic diseases, especially cancer and CVDs. However, although many clinical trials have been conducted with vitamins (E, C or their combinations) their in vivo protective effect remains uncertain. Therefore the possibility that the complex mixture of phytochemicals in foods may contribute to their protecting effects has been raised. In this concept, it is possible multiple compounds to act through complimentary or synergistic mechanisms to present a greater biologic effect than can be achieved by any individual component To investigate this hypothesis, a double-blind, randomized, and placebo-controlled clinical trial was conducted in order to investigate the effects of a multi-micronutrient supplement against oxidative stress in apparently healthy adults.

DETAILED DESCRIPTION:
This was a double-blind, block randomized, parallel-arm, placebo-controlled, eight-week study. Initially 77 apparently healthy volunteers were recruited to participate in the study. 62 volunteers were enrolled in the study and assigned to either the MM group (n = 32) or the placebo group (n = 30) using a stratified randomization to guarantee comparability of age, sex and BMI distribution between the two groups. The randomization code was prepared by a staff member who was not involved in running the trial, by using computer-generated random numbers. At the initiation of the study, the subjects received 5 bottles (0.5L each) of the MM or placebo, which were made indistinguishable by their identical packaging. At 4 weeks the subjects received again 5 bottles. The subjects were asked to consume 80mL per day, preferably after meals. The dose was chosen based on the commercially recommended level. At each visit, the remaining volume of the supplement was counted by research coordinators. The subjects were excluded from the analysis if they consumed <80% of the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI: 23-30

Exclusion Criteria:

* regular use of dietary supplements or medications
* being on slimming or any other special diet
* hypertension
* metabolic or endocrine disease
* gastrointestinal disorders
* recent history of medical or surgical events

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of isoprostane levels at 4 weeks | 0, 4 weeks
  urinary isoprostane
Change from Baseline of isoprostane levels at 8 weeks | 0, 8 weeks
  urinary isoprostane
Change from Baseline of DNA/RNA damage at 4 weeks | 0, 4 weeks
  urinary DNA/RNA damage
Change from Baseline of DNA/RNA damage at 8 weeks | 0, 8 weeks
  urinary DNA/RNA damage
Change from Baseline of protein carbonyls levels at 4 weeks | 0, 4 weeks
  serum
Change from Baseline of protein carbonyls levels at 8 weeks | 0, 8 weeks
  serum
Change from Baseline of oxLDL levels at 4 weeks | 0, 4 weeks
  serum
Change from Baseline of oxLDL levels at 8 weeks | 0, 8 weeks
  serum
Change from Baseline of TBARS levels at 4 weeks | 0, 4 weeks
  serum
Change from Baseline of TBARS levels at 8 weeks | 0, 8 weeks
  serum
Change from Baseline of serum resistant in oxidation at 4 weeks | 0, 4 weeks
  ex vivo serum oxidation with cupper
Change from Baseline of serum resistant in oxidation at 8 weeks | 0, 8 weeks
  ex vivo serum oxidation with cupper
Change from Baseline of anti-oxidant enzymes activity at 4 weeks | 0, 4 weeks
  serum
Change from Baseline of anti-oxidant enzymes activity at 8 weeks | 0, 8 weeks
  serum

SECONDARY OUTCOMES:
Change from Baseline of Platelet aggregation against PAF at 4 weeks | 0, 4 weeks
  PRP aggregation against PAF
Change from Baseline of Platelet aggregation against PAF at 8 weeks | 0, 8 weeks
  PRP aggregation against PAF
Change from Baseline of Platelet aggregation at against ADP 4 weeks | 0, 4 weeks
  PRP aggregation against ADP
Change from Baseline of Platelet aggregation against ADP at 8 weeks | 0, 8 weeks
  PRP aggregation against ADP
Change from Baseline of Platelet aggregation against TRAP at 4 weeks | 0, 4 weeks
  PRP aggregation against TRAP
Change from Baseline of Platelet aggregation against TRAP at 8 weeks | 0,8 weeks
  PRP aggregation against TRAP
Change from Baseline of Inflammatory markers at 4 weeks | 0, 4 weeks
  serum LpPLA2 activity
Change from Baseline of Inflammatory markers at 8 weeks | 0,8 weeks
  serum LpPLA2 activity

REFERENCES:
- [Derived] Fragopoulou E, Gavriil L, Argyrou C, Malagaris I, Choleva M, Antonopoulou S, Afxentiou G, Nikolaou E. Suppression of DNA/RNA and protein oxidation by dietary supplement which contains plant extracts and vitamins: a randomized, double-blind, placebo-controlled trial. Lipids Health Dis. 2018 Aug 16;17(1):187. doi: 10.1186/s12944-018-0836-z. PMID 30115068